CLINICAL TRIAL: NCT00836654
Title: Two-Arm, Randomized (2:1), Open-Label Phase II/III Study in EpCAM Positive Cancer Patients With Symptomatic Malignant Ascites Using the Trifuncitonal Bispecific Antibody Removab (Anti-EpCAM x Anti-CD3) Versus an Untreated Control Group
Brief Title: Study in EpCAM Positive Patients With Symptomatic Malignant Ascites Using Removab Versus an Untreated Control Group
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Neovii Biotech (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 60117
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Last update posted 2009-02-05 (Estimated); Status verified 2009-02

CONDITIONS: EpCam Positive Tumor (e.g.Ovarian, Gastric, Colon, Breast); Malignant Ascites
Keywords: EpCAM positive tumor; malignant ascites; intraperitoneal
MeSH Terms: interventions — catumaxomab; Paracentesis

ARMS (2):
- 1 Catumaxomab (Active Comparator): Patient received Catumaxomab and paracentesis
  Interventions: Biological: Catumaxomab (Removab); Procedure: paracentesis
- 2: (No Intervention): Patient treated by paracentesis alone, but after the second paracentesis the patient is able to cross-over in the Catumaxomab-arm

INTERVENTIONS:
Biological: Catumaxomab (Removab) — Puncture free survival
  Other Names: Removab
  Arms: 1 Catumaxomab
Procedure: paracentesis
  Arms: 1 Catumaxomab

SUMMARY:
The study will be performed to obtain further efficacy and safety data in order to obtain a marketing authorization (pivotal study). In addition, health economic data are to be collected.

ELIGIBILITY:
Inclusion Criteria:

* histological confirmed diagnosis cancer
* symptomatic malignant ascites
* EpCAM positive tumor
* EOCG 0-2
* negative pregnancy

Exclusion Criteria:

* acute or chronic infection
* exposure to investigational product, cancer chemo- or radiotherapy within the last 28 days
* previous treatment with mouse monoclonal antibodies
* known or suspected hypersensitivity to Removab or similar antibodies
* inadequate renal function
* inadequate hepatic function (AST, ALt, GTP,< x ULN; bilirubin <1.5xULN)
* Platelets > 80000 cells/mm3; absolute neutrophil count (ANC) < 1500 cells/mm3
* BMI < 17
* Patients with reduced nutritional status
* Ileus within the last 30 days
* Brain metastases in cancer history
* Pregnant and nursing women
* history of myocardial infarction, congestive heart failure or relevant cardiac arrhythmia within previous 3 months
* inadequate respiratory function in option of investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2004-09; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

REFERENCES:
- [Background] Ruf P, Lindhofer H. Induction of a long-lasting antitumor immunity by a trifunctional bispecific antibody. Blood. 2001 Oct 15;98(8):2526-34. doi: 10.1182/blood.v98.8.2526. PMID 11588051
- [Background] Riesenberg R, Buchner A, Pohla H, Lindhofer H. Lysis of prostate carcinoma cells by trifunctional bispecific antibodies (alpha EpCAM x alpha CD3). J Histochem Cytochem. 2001 Jul;49(7):911-7. doi: 10.1177/002215540104900711. PMID 11410615
- [Background] Zeidler R, Mysliwietz J, Csanady M, Walz A, Ziegler I, Schmitt B, Wollenberg B, Lindhofer H. The Fc-region of a new class of intact bispecific antibody mediates activation of accessory cells and NK cells and induces direct phagocytosis of tumour cells. Br J Cancer. 2000 Jul;83(2):261-6. doi: 10.1054/bjoc.2000.1237. PMID 10901380
- [Background] Zeidler R, Reisbach G, Wollenberg B, Lang S, Chaubal S, Schmitt B, Lindhofer H. Simultaneous activation of T cells and accessory cells by a new class of intact bispecific antibody results in efficient tumor cell killing. J Immunol. 1999 Aug 1;163(3):1246-52. PMID 10415020
- [Background] Heiss MM, Strohlein MA, Jager M, Kimmig R, Burges A, Schoberth A, Jauch KW, Schildberg FW, Lindhofer H. Immunotherapy of malignant ascites with trifunctional antibodies. Int J Cancer. 2005 Nov 10;117(3):435-43. doi: 10.1002/ijc.21165. PMID 15906359
- [Derived] Wimberger P, Gilet H, Gonschior AK, Heiss MM, Moehler M, Oskay-Oezcelik G, Al-Batran SE, Schmalfeldt B, Schmittel A, Schulze E, Parsons SL. Deterioration in quality of life (QoL) in patients with malignant ascites: results from a phase II/III study comparing paracentesis plus catumaxomab with paracentesis alone. Ann Oncol. 2012 Aug;23(8):1979-1985. doi: 10.1093/annonc/mds178. Epub 2012 Jun 24. PMID 22734013